CLINICAL TRIAL: NCT04527172
Title: Neuromuscular Ultrasonography Utility for Detection of Peripheral Neuropathy in Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira M elSonbaty, Principal Investigator, Assiut University
Other Study IDs: 17200346
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Neuropathy; System; Lupus Erythematosus
Keywords: Neuromuscular ultrasound; SLE; Peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Lupus Erythematosus, Systemic | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- systemic lupus patients: Nerve conduction study and neuromuscular ultrasound for median , ulnar, tibial, peroneal and sural nerves
  Interventions: Diagnostic Test: neuromuscular ultrasound
- Healthy subjects: Nerve conduction study and neuromuscular ultrasound for median , ulnar, tibial, peroneal and sural nerves
  Interventions: Diagnostic Test: neuromuscular ultrasound

INTERVENTIONS:
Diagnostic Test: neuromuscular ultrasound — ultrasound to visualize the peripheral nerves of lupus patients and to compare it with results of the raditional electrophysiological studies
  Other Names: nerve conduction study

SUMMARY:
This study aims to evaluate the rule of NMUS in detection of peripheral neuropathy in SLE patient and to correlate it to traditional neurophysiological studies, clinical signs and activity of SLE.

DETAILED DESCRIPTION:
The frequency of SLE peripheral neuropathy documented by electrophysiology has been estimated to be approximately 30%.

The term peripheral neuropathies include symmetric polyneuropathy, single and multiple mononeuropathy, and radiculopathy.

There has been increasing interest in using ultrasonography (US) to aid peripheral neuropathy diagnosis and studies have shown good correlation with other imaging modalities. US is a non-invasive and inexpensive imaging device that has become widely available as a diagnostic tool at many fields.

so systemic lupus patients were enrolled in the study , performed nerve conduction study and neuromuscular ultrasound for bil. median, ulnar, peroneal, tibial and sural nerves , on statistics the cross sections were compared in neurophusiologically affected and non affected nerves, also the sensitivity and specifity of NMUS in comparison to the traditional NCS was calculated

ELIGIBILITY:
Inclusion Criteria:

1. All adult SLE patients who was admitted to Rheumatology & Rehabilitation department of Assuit university hospital during time frame of study.
2. apparently healthy subjects with normal electrophysiological study
3. verbal consent, free and informed

Exclusion Criteria:

* • Other causes of peripheral neuropathy:

  1. Traumatic
  2. Purely degenerative
  3. Diabetic
  4. Toxic
  5. Infections
  6. Drug induced

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All adult SLE patientA who was admitted to Rheumatology & Rehabilitation department of Assuit university hospital during time frame of study. and apparently healthy subjects with normal electrophysiological study
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
evaluate the rule of NMUS in detection of peripheral neuropathy in SLE patient | 6months
  Measuring sensitivity and specificity of neuromuscular ultrasound in comparison to nerve conduction study
Describing the patterns of peripheral nerve affection in SLE patient | 6months
  Evaluating different studied nerves clinically, electrophyiologically and by neuromuscular ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Tayseer Khedr, PHD, Study Director — Assiut University
Locations (1):
- Assuit university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the priciple investigator only will know the results of neurophysiology done to the patients then the images were furtherly evaluated (offline) by another expert rheumatologist who was blinded to both clinical and electrophysiological data of the patients. Any conflict in reporting was refered to a third expert rheumatologist to put the final decision.

REFERENCES:
- [Derived] Mahran SA, Galluccio F, Khedr TM, Elsonbaty A, Allam AE, Garcia Martos A, Osman DMM, Matucci-Cerinic M, Guiducci S, Galal MAA. Peripheral neuropathy in systemic lupus erythematosus: what can neuromuscular ultrasonography (NMUS) tell us? A cross-sectional study. Lupus Sci Med. 2021 Jul;8(1):e000521. doi: 10.1136/lupus-2021-000521. PMID 34312211